CLINICAL TRIAL: NCT04659304
Title: A Multi-Center , Sequential Dose Escalation Study, Evaluating Safety and Tolerability of Allocetra-OTS in Patients With COVID-19
Brief Title: Study Evaluating Safety and Tolerability of Allocetra-OTS in Patients With COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENX-CL-03-001
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Cell therapy; Allocetra-OTS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: sequential dose escalation using a 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): Single Intravenous (IV) dose of Allocetra-OTS with 5x10^9 cells
  Interventions: Drug: Allocetra-OTS
- Cohort 2 (Active Comparator): Single Intravenous (IV) dose of Allocetra-OTS with 10x10^9 cells
  Interventions: Drug: Allocetra-OTS
- Cohort 3 (Active Comparator): Two IV doses of Allocetra-OTS with 10x10^9 cells in each dose
  Interventions: Drug: Allocetra-OTS

INTERVENTIONS:
Drug: Allocetra-OTS — Cell-based therapy comprised of allogeneic non-HLA matched peripheral blood mononuclear cells induced to an early apoptotic state.

SUMMARY:
Phase 1b, multi-center, open label, sequential dose escalation trial assessing 3 dose cohorts using a 3+3 design to evaluate safety and tolerability of Allocetra-OTS in adult patients with moderate COVID-19. The sample size for this trial is anticipated to range from 9 to 18 patients.

DETAILED DESCRIPTION:
Potential patients, who will be identified as suffering from moderate COVID-19 (as set forth in the FDA guidance for industry dated May 2020) will be recruited.

After the patient has signed the Informed Consent Form (ICF), and after confirmation that the patient meets all eligibility criteria, the patient will be enrolled to the relevant dose group according to the following sequential design:

Single Intravenous (IV) dose of Allocetra-OTS with 5x10^9 cells, Single Intravenous (IV) dose of Allocetra-OTS with 10x10^9 cells, Two IV doses of Allocetra-OTS with10x10^9 cells each dose (separated by 72 hours).

Each dose cohort will consist of 3 and up to 6 patients. In each dose cohort, starting with dose cohort 1, a single patient will be enrolled and dosed. If no dose limiting toxicity (DLT) is observed after at least 1 week and following review of relevant safety data of the first patient in that cohort by the DMC, 2 additional patients will be enrolled.

If no DLT is seen in the initial 3 dosed patients within a certain cohort and following DMC review, the first patient in the next dose cohort can be enrolled, repeating the same sequence of enrollment as described above.

If 1 DLT is seen in the initial 3 dosed patients within a certain cohort, the cohort will be expanded to a total of 6 patients. If >2/6 patients experience a DLT, the MTD will be reached. If no more than 1 patient out of 6 experiences a DLT, the next sequence of enrollment will be continued.

DMC will review and assess safety data at the predefined timepoints to recommend on cohort expansion or cohort escalation.

Investigational Product (IP) administration will occur on Day 1 within 12±4 hours from the time of eligibility.

Following IP administration (Day 1), patients will be followed for safety and efficacy assessments through 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female > 18 and < 80 years of age.
2. Laboratory confirmation of SARS-CoV-2 infection by RT-PCR from any diagnostic sampling source.
3. Patient hospitalized due to COVID-19 in the last 24 hours.
4. Hospitalized patients meeting the criteria for moderate COVID-19, as set forth by the May 2020 FDA Guidance for Industry: COVID-19: Developing Drugs and Biological Products for Treatment or Prevention, Patients with symptoms of moderate illness with COVID-19, which could include any symptom of mild illness (such as fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea) or shortness of breath with exertion with at least one of the following clinical signs:

   1. Respiratory rate: ≥ 20 breaths/minute;
   2. SpO2: > 93% on room air at sea level;
   3. Heart rate: ≥ 90 beats/minute;
5. Signed written informed consent by the patient.
6. Women and men who are of childbearing potential, willing to use acceptable contraceptive measures during 4 weeks from enrolment .

Exclusion Criteria:

1. Any signs indicative of Severe or Critical Illness Severity requiring hospitalization as defined below:

   Severe COVID-19: Shortness of breath in rest, or respiratory distress, or respiratory rate (RR≥30 per minute , or heart rate (HR) ≥125 bpm, or SpO2≤93% on room air at sea level or PaO2/FiO2<300

   Critical COVID-19- at least one of the following:
   * Respiratory failure required at least one of the following: mechanical ventilation, oxygen delivered by high-flow nasal cannula, noninvasive positive pressure ventilation, ECMO.
   * Shock
   * Multi-organ dysfunction/failure.
2. Women who are pregnant or breast feeding.
3. Weight <50 kg or >110 kg.
4. Stage 4 and 5 severe chronic kidney disease or requiring dialysis with eGFR < 30 ml/min.
5. Patients with active malignant tumor.
6. Patients who are participating in other concurrent investigational clinical trials or have been treated with any experimental agents within 30 days prior to enrollment.
7. Known active chronic viral infections including, but not limited to, active HBV, HCV, or HIV/AIDS or other chronic infections.

   Based on medical history and concomitant therapies that would suggest infection, have suspected clinical diagnosis of current active TB or, if known, latent TB treated for less than 4 weeks with appropriate anti-TB therapy per institutional guidelines; Based on medical history and concomitant therapies that would suggest infection, suspected serious, active bacterial, fungal, viral (including, but not limited to, active HBV, HCV, or HIV/AIDS).
8. Known immunocompromised state or immunosuppressing medications taken for indications other than SARS-CoV-2 (i.e., agents including chronic corticosteroids > 10 mg/day, azathioprine, cyclosporine, cyclophosphamide).
9. Known New York Heart Association (NYHA) class III and IV heart failure or unstable angina, ventricular arrhythmias, active ischemic heart disease , or myocardial infarction within six months prior to diagnosis of COVID-19.
10. Known active upper gastrointestinal (GI) tract ulceration or hepatic dysfunction including but not limited to biopsy-proven cirrhosis; end-stage cirrhosis (Child Pugh Class C); portal hypertension; episodes of past upper GI bleeding attributed to portal hypertension; or prior episodes of hepatic failure, encephalopathy, or coma.
11. Patients with Glasgow Coma Scale (GCS) <13 with verbal score <5.
12. Estimated GFR < 25 ml/min.
13. Hemoglobin < 8 gr%.
14. Patients with history of chronic liver disease, evidence of acute cholangitis or cholecystitis. Patients with at least one of the following:

    * ALT or AST > 5X ULN (upper limit of normal range)
    * Bilirubin > 3 X ULN
    * Combination of ALT/AST > 3 X ULN and elevated direct bilirubin>ULN
15. Known history of transfusion reactions, hemolytic anemia, or allergic reaction.
16. Organ allograft or previous history of stem cell transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | 28 days
  Number and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs).
Maximum Tolerated Dose (MTD) | 28 days
  The highest dose of Allocetra-OTS that did not cause a Dose-Limiting Toxicity (DLT) in 2/6 cohort patientsor maximally administered dose if no DLT is seen.

SECONDARY OUTCOMES:
Efficacy - PaO2 or SO2/FiO2 Ratio | 28 days
  Change in PaO2 or SO2/FiO2 Ratio
Efficacy - mortality | 28 days
  All-cause mortality
Efficacy - organ function / support measurements | 28 days
  Oxygen free days, vasopressors free days, cumulative days in ICU or IMU
Efficacy - NEWS2 Score | 28 days
  Change from baseline in National Early Warning Score 2 (NEWS2)

CONTACTS AND LOCATIONS:
Overall Officials: Oren Hershkovitz, PhD, Study Director — Enlivex Therapeutics R&D

IPD SHARING:
Plan to Share IPD: No
Patient data will not contain any information which would make the patient identifiable. Data will be processes and shared using patient study number only.